CLINICAL TRIAL: NCT06291324
Title: Wearable Activity Tracker Devices and Cancer-Related Fatigue: A Clinical Utility Pilot Study For Patients Undergoing Anti-Cancer Treatment
Brief Title: WATD and Cancer-Related Fatigue: A Study For Patients Undergoing Anti-Cancer Treatment
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00103472; LCI-SUPP-CRF-WATD-001 (Other: Atrium Health); NCI-2024-06147 (Other: National Cancer Institute)
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Breast Cancer
Keywords: Fatigue
MeSH Terms: conditions — Pancreatic Neoplasms; Breast Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the feasibility of using a commercial WATD (Wearable Activity Tracker Device) to collect HRV (Heart Rate Variability) data from pancreatic and breast cancer patients.

DETAILED DESCRIPTION:
This feasibility study is designed to evaluate the collection of longitudinal HRV (Heart Rate Variability) data and assess acceptability of the device among adult cancer patients in the research setting. Over the course of the four-week study, participants will be asked to provide experiential diaries detailing adherence to and acceptability of the WATD (Wearable Activity Tracker Device) and conduct PRO (Patient Reported Outcome) measures at week two and week four (end of study). During the final research visit at week four, subjects will return the WATD and will complete the acceptability survey. Each week of the four-week study, the WATD data and experiential diaries will be downloaded for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information
* Patients pancreatic or invasive breast cancer per enrolling investigator who is planning on or has started anti-cancer treatment. Note: Patients with cancer who are not planning to receive anti-cancer treatment are not eligible for study participation
* Patients with any severity of self-reported fatigue per enrolling investigator
* Age ≥ 18 years at the time of consent
* Ability to read and understand the English language
* As determined by the enrolling investigator, the ability of the participant to understand and comply with study procedures (i.e., completing questionnaires and device return) for the entire length of the study

Exclusion Criteria:

* Any documented, clinically significant cardiac-related abnormality per enrolling investigator that could compromise the outcome of the study. NOTE: The heart rate data collected using the WATD will not be used for patient care.
* Other factors or conditions, per investigator discretion, for which participation in the study would not be in the patient's best interest or could interfere with study assessment results or preclude study completion
* No internet, Wi-Fi access or email account
* No access to a smartphone or mobile device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years of age who have any stage pancreatic or breast cancer per enrolling investigator and have self-reported fatigue
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Adherence and acceptability | Day 14
  Adherence is a binary variable and will be determined based on whether the participant uploads HRV data each morning at least 75% of the days during the 14-day trial. Acceptability is a binary variable, and it is based on participant's response to the question whether they find the Wearable Activity Tracker Device (WATD) easy to use in the acceptability survey.

SECONDARY OUTCOMES:
Theme | Day 14
  Themes are categories of consolidated meaning derived from qualitative data that concern acceptability and adherence to using the Wearable Activity Tracker Device (WATD). They are derived based on qualitative analysis of the Experiential Diary, Acceptability survey open-ended data, and lifestyle behavior data. Theme is a categorical variable.
Heart rate variability (HRV) | Day 14
  HRV is the variation in the time intervals between adjacent heartbeats. It is a continuous variable and is measured by the Wearable Activity Tracker Device (WATD).

CONTACTS AND LOCATIONS:
Overall Officials: Dori Beeler, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No